CLINICAL TRIAL: NCT03031366
Title: A Novel Approach for Transjugular Intrahepatic Portocaval Shunt Creation Using Real-time Three Dimensional Roadmap
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, luo xuefeng, attending doctor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3D roadmap for TIPS
Record Dates: First submitted 2017-01-21; First posted 2017-01-25 (Estimated); Last update posted 2019-01-08 (Actual); Status verified 2019-01

CONDITIONS: Portal Hypertension
MeSH Terms: conditions — Hypertension, Portal

STUDY DESIGN:
Intervention Model Description: TIPS creation using real-time 3D roadmap
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3D roadmap (Experimental): TIPS was established using 3d roadmap guidance
  Interventions: Other: 3d roadmap guidance
- conventional TIPS (Active Comparator): conventional TIPS procedure using wedged hepatic venography
  Interventions: Other: conventional TIPS procedure

INTERVENTIONS:
Other: 3d roadmap guidance — TIPS was established using 3d roadmap
  Arms: 3D roadmap
Other: conventional TIPS procedure — conventional TIPS procedure using wedged hepatic venography
  Arms: conventional TIPS

SUMMARY:
TIPS creation has been widely used to treat the complications associated with portal hypertension. In association with increased operator experience and the ongoing development of imaging modalities, the rate of major complications associated with TIPS has decreased significantly in the past decades. However, the passage of a curved needle from the hepatic vein into the portal vein still remains a challenging and time-consuming part of the procedure and is associated with puncture-related complications that are potentially fatal.Three-dimensional roadmap guidance has been widely applied in various interventions. The aim of the present study is to prospectively assess the feasibility and efficacy of real-time 3D roadmap guidance during TIPS creation.

ELIGIBILITY:
Inclusion Criteria:

cirrhosis complications of portal hypertension requiring TIPS

Exclusion Criteria:

non-cirrhotic portal hypertension complete occlusion of intrahepatic portal vein gastro-renal shunt presence of liver tumor pregnancy other contradictions of TIPS

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-02-13 (Actual); Primary Completion 2017-05-30 (Actual); Study Completion 2017-05-30 (Actual)

PRIMARY OUTCOMES:
Technical success rate | 1 month
  number of patients who have received TIPS creation technically successfully
number of punctures | 1 month
  number of intrahepatic punctures for TIPS creation

SECONDARY OUTCOMES:
radiographic fluoroscopy time for portal vein entry | 1 month
  duration of radiographic fluoroscopy for portal vein entry
radiographic fluoroscopy time for the whole procedure | 1 month
  duration of radiographic fluoroscopy for the whole procedure
procedural time | 1 month
  procedural time

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided